CLINICAL TRIAL: NCT04216680
Title: Asthma and Intimate Partner Violence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Jewish Health (Other)
Responsible Party: Principal Investigator, Eileen Wang, Assistant Professor, National Jewish Health
Other Study IDs: HS-3068
Record Dates: First submitted 2019-12-31; First posted 2020-01-03 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Asthma; Domestic Violence
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a cross-sectional observational study on adult asthmatics evaluating the relationship between asthma control and psychosocial factors to include intimate partner violence, stress, anxiety, depression, post-traumatic stress disorder.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma as defined as postbronchodilator response of at least 12% and 200 milliliters improvement in forced expiratory volume in 1 second (FEV1) or forced vital capacity and/or evidence of positive airway hyperresponsiveness.

Exclusion Criteria:

* Medical factors that would preclude participation as determined by the investigators. Examples include blindness, mental illness that grossly impairs judgment, or active injury requiring treatment.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult asthmatics ages 18-69 years who are able to participate in a questionnaire-based study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-01-02 (Estimated); Primary Completion 2021-01-02 (Estimated); Study Completion 2021-01-02 (Estimated)

PRIMARY OUTCOMES:
Asthma Control Test | last 30 days
  asthma control scored on scale of 0-25 with higher numbers reflecting better control.

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States